CLINICAL TRIAL: NCT00828269
Title: Evaluation of RNA Quality and the Reproducibility of Gene Expression Profiling From Liver Tissue Obtained by Fine Needle Aspiration in Patients With Chronic Hepatitis C.
Brief Title: Evaluation of RNA From the Liver Tissue Obtained in Patients With Chronic Hepatitis C (0000-123)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0000-123; 123; 2009_518
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Hepatitis C
Keywords: Patients with Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- 1 (No Intervention): Liver tissue biopsy
  Interventions: Procedure: Comparator: Fine needle aspiration biopsy

INTERVENTIONS:
Procedure: Comparator: Fine needle aspiration biopsy — Visit 1: Screening Visit 2 (7-14 days from screening): Core needle biopsy and fine needle aspiration biopsy - liver.
  Visit 3:(7 days from visit 2): Fine needle aspiration biopsy - liver. Visit 4: (14 days from Visit 3): follow-up visit

SUMMARY:
The purpose of this study is to evaluate the quality of the RNA and the reproducibility of gene expression profiling from liver tissue samples obtained by fine needle aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic hepatitis C (Genotype 1)
* Patient has the ability to avoid use of anticoagulants, nonsteroidal anti-inflammatory drugs and aspirin for at least 5 days before the liver biopsy

Exclusion Criteria:

* Patient has received any approved or investigational drugs for the treatment of hepatitis C in the six months before the liver biopsy
* Patient has HIV or Hepatitis B virus
* Patient has been diagnosed with liver cancer
* Patient has evidence of cirrhosis on any previous liver biopsy
* Patient has confirmed alcohol abuse in the last 12 months
* Patient has participated in any investigational drug study within 90 days before the current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the probability that fine needle aspiration of the liver results in RNA suitable to conduct gene expression tests. | 5 weeks

SECONDARY OUTCOMES:
Comparison of qPCR and microarray signature from patients with no or minimal fibrosis to that from patients with moderate to advanced fibrosis. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC